CLINICAL TRIAL: NCT02776189
Title: Comparative Study of Dexmedetomidine-midazolam Combination and Propofol-midazolam Combination for MRI Brain in Paediatric Patient
Brief Title: Dexmedetomidine Verses Propofol for Paediatric MRI Brain
Acronym: DPMP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maharashtra University of Health Sciences (Other)
Responsible Party: Principal Investigator, Nazmeen Sayed, Assistant Professor, Department of Anaesthesia, Lokmanya Tilak Municipal Medical College and Hospital, Maharashtra University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: iec/30/12
Record Dates: First submitted 2016-05-11; First posted 2016-05-18 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Brain Diseases
Keywords: Anaesthesia; MRI; Brain
MeSH Terms: conditions — Brain Diseases | interventions — Dexmedetomidine; Propofol; Midazolam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Midazolam & Dexmedetomidine (Experimental): Intra nasal midazolam 0.2 mg per kg body weight before intravenous canulation. Intravenous dexmedetomidine 1 mcg per kg body weight over 10 minutes followed by infusion of dexmedetomidine at dose of 1 mcg per kg body weight per hour till end of procedure
  Interventions: Drug: Dexmedetomidine; Drug: Midazolam
- Midazolam & Propofol (Active Comparator): Intra nasal midazolam 0.2 mg per kg body weight before intravenous canulation. Intravenous propofol 2 mg per kg body weight followed by infusion of propofol at a dose of 100 mcg per kg body weight per min till end of procedure
  Interventions: Drug: propofol; Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — intravenous dexmedetomidine 1 mcg per kg body weight over 10 minutes followed by infusion of dexmedetomidine at dose of 1 mcg per kg body weight per hour till end of procedure
  Other Names: Dexem
  Arms: Midazolam & Dexmedetomidine
Drug: propofol — intravenous propofol 2mg per kg body weight followed by infusion of propofol at a dose of 100 mcg per kg body weight per min till end of procedure
  Other Names: propoven; diprivan
  Arms: Midazolam & Propofol
Drug: Midazolam — Intra nasal midazolam 0.2 mg per kg body weight before intravenous canulation
  Other Names: Versed; Fulsed

SUMMARY:
MRI though not painful requires deep sedation for children due to the loud noise created. With deep sedation comes respiratory depression so the interest in Dexmedetomidine. For standardization MRI brain was chosen and also for the fact that patients usually have history of convulsions where drugs like ketamine may not be a good option. Patients were recruited after ethics committee approval. After pre-medication with intranasal midazolam 0.2 mg/kg body weight, Intravenous access was established and then patients were divided in two groups. One group received intravenous propofol 2mg/Kg and infusion of 100mcg/per kg body weight per minute. The other group received intravenous bolus of Dexmedetomidine 1mcg/kg over 10 minutes and then a infusion of Dexmedetomidine 1mcg/kg/hour.

Primary out come was to study the recovery time of patients sedated with Dexmedetomidine compared to patients sedated with propofol for paediatric MRI brain. Secondary outcome were analysed in terms of time for induction,procedural disruptions due to awakening and haemodynamic stability . Follow up was done on phone for any adverse events.

DETAILED DESCRIPTION:
Patients were evaluated on out patient department basis. On the day of MRI nil per oral status of 6 hours was confirmed and consent taken from the parent. In recovery room after recording of vitals, children were given intranasal midazolam 0.2mg/kg body weight. The intravenous line was secured after the child was sedated. Patients were then divided in two groups. In the MRI console, the dexmedetomidine group received intravenous dexmedetomidine 1mcg/kg body weight over 10 minutes. An intravenous infusion of dexmedetomidine was then started at 1mcg/kg/hour.

The propofol group received 2mg /kg of intravenous propofol and an infusion of 100mcg/kg/minute.

MRI monitoring included pulseoximetry, cardioscope, respiratory pattern and rate. Oxygen was delivered by nasal prongs. Primary outcome measured was the time for recovery.

Secondary outcomes were number of awakening during procedure, haemodynamic stability, induction time and any adverse events.

After MRI the children were observed in the recovery room and discharged after achieving 'modified aldred score' of 10. Vitals and any adverse events were recorded during this phase.

ELIGIBILITY:
Inclusion Criteria:

* children posted for elective MRI brain
* American society of anaesthesiologist physical status I and II

Exclusion Criteria:

* age less than 1 year and more than 7 years
* American society of anaesthesiologist physical status III and IV
* emergency cases
* upper respiratory tract infection
* patients on digoxin and beta blockers
* allergy to study drugs
* Body mass index more than 35

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2012-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Recovery time | 4 hours after procedure
  Recovery time - time from the end of the procedure till the patient achieves a Modified aldred score of 10.Modified Aldred Score- a score from 0- 10 considering 5 parameters of activity, oxygen saturation, respiration, circulation and consciousness each given score 0,1,2. Score of 10 patients can be sent home after outpatient anaesthesia.

SECONDARY OUTCOMES:
Time for induction | One hour
  time for induction - time from administration of drug to the patient till the patient is sedated enough for allowing positioning for MRI
Procedural disruptions due to awakening of the patient | one hour
  Number of patients in each group who had one or more awakening during the procedure was compared
Bradycardia | 6 hours
  number of patients having bradycardia after induction till recovery was compared. Bradycardia is heart rate less than 60 beats per minute
Desaturation | 6 hours
  Number of patients in each group that had desaturation was compared. Desaturation was defined as drop in oxygen saturation of less than 98 percent inspite of supplemented oxygen. Normal oxygen saturation as measured by pulse oximeter is 100 percent on room air.

CONTACTS AND LOCATIONS:
Overall Officials: nazmeen I Sayed, MBBS,DNB, Principal Investigator — Lokmanya Tilak Municipal Medical College and Hospital; Naina Dalvi, MBBS,MD, Principal Investigator — Lokmanya Tilak Municipal Medical College and Hospital
Locations (1):
- Lokmanya Tilak Municipal General Hospital and Lokmanya Tilak Municipal Medical College, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Yes